CLINICAL TRIAL: NCT00670592
Title: A Phase IA/II, Multi-center, Open-label Study of HCD122 Administered Intravenously Once Weekly for Four Weeks in Adult Patients With Advanced Non-Hodgkin's or Hodgkin's Lymphoma Who Have Progressed After at Least Two Prior Therapies (CHIR-12.12-LYM-01)
Brief Title: Study of HCD122 in Adults With Non-Hodgkin's or Hodgkin's Lymphoma Who Have Progressed After at Least Two Prior Therapies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHCD122A2103; 2007-004888-22 (EudraCT Number)
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2014-01

CONDITIONS: Non-Hodgkin's Lymphoma; Hodgkin's Lymphoma
Keywords: HCD122; CD40; NHL; HL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — lucatumumab

ARMS (1):
- HCD122 (Other)
  Interventions: Drug: HCD122

INTERVENTIONS:
Drug: HCD122

SUMMARY:
This study is to evaluate the highest tolerated dose, safety and activity of HCD122 in adults with non-Hodgkin's or Hodgkin's lymphoma who have received at least two prior therapies.

ELIGIBILITY:
Inclusion criteria:

Patients may be included in the study if they meet all of the following criteria:

* Patients must have confirmed diagnosis of HL or NHL (follicular, marginal zone / MALT, diffuse large B-cell, or mantle cell) per REAL/WHO classification
* Patients must have progressed after at least 2 prior therapies (autologous stem cell transplantation is considered as 1 therapy)
* Patients must be ≥ 18 years
* Patients must have life expectancy > 3 months
* Patient must have adequate laboratory results
* Patients must have WHO Performance Status grade 0, 1, or 2
* Patients must have at least one site of measurable disease
* Patients must have discontinued any previous monoclonal antibody or radioimmunotherapy, and must have recovered fully from the side effects of that treatment prior to beginning study treatment.
* Patients must be willing and able to sign the informed consent form and comply with the study protocol

Exclusion criteria:

Patients will be excluded from the study if they meet any of the following criteria:

* Patients who have been treated with any anti-CD40 antibody
* Patients who have received prior allogeneic stem cell transplant
* Patients who have had a prior anaphylactic or other severe infusion reaction such that the patient is unable to tolerate human immunoglobulin or monoclonal antibody administration
* Patients who have history or clinical evidence of central nervous system, meningeal, or epidural disease including brain metastasis
* Women of child-bearing potential (WCBP) who are pregnant or breast feeding.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2008-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Primary endpoints (phase I) - Incidence rate of DLT and AE | 2 years
Primary endpoint (phase II) - Response rate | 2 years

SECONDARY OUTCOMES:
Adverse events by frequency, severity, and duration; pharmacokinetics; immunogenicity; response duration; time to progression | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticlas, Study Director — Novartis Pharmaceuticals
Locations (28):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - St. Francis Cancer Research Foundation Dept.ofSt.FrancisCancerRes.(2), Beech Grove, Indiana
  - Dana Farber Cancer Institute SC-5, Boston, Massachusetts
  - Wake Forest University Baptist Medical Center Dept. of Industry Research (2), Winston-Salem, North Carolina
  - University of Texas/MD Anderson Cancer Center Dept.ofMDAndersonCancerCtr(3), Houston, Texas
- Australia (2):
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Prahran, Victoria
- Belgium (3):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Godinne
  - Novartis Investigative Site, Leuven
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (6):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Benite Cédex
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (3):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pisa, PI
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, Korea, South Korea
- United Kingdom (2):
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London

REFERENCES:
- See also: Results for CHCD122A2103 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=10903